CLINICAL TRIAL: NCT02442557
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and T-cell Tolerizing Effect of DC-TAB in Healthy Volunteers
Brief Title: Safety and Dose-finding Study of DC-TAB in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Delta Crystallon BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DC-001
Record Dates: First submitted 2015-05-01; First posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Multiple Sclerosis
Keywords: alpha B-crystallin; immune tolerance
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- single dose 4 mg (Active Comparator): a single intravenous injection of 4 mg DC-TAB
  Interventions: Biological: recombinant human alpha B-crystallin
- single dose 12.5 mg (Active Comparator): a single intravenous injection of 12.5 mg DC-TAB
  Interventions: Biological: recombinant human alpha B-crystallin
- single dose 25 mg (Active Comparator): a single intravenous injection of 25 mg DC-TAB
  Interventions: Biological: recombinant human alpha B-crystallin
- single dose 37.5 mg (Active Comparator): a single intravenous injection of 4 mg DC-TAB
  Interventions: Biological: recombinant human alpha B-crystallin
- single dose placebo (Placebo Comparator): a single intravenous injection of placebo
  Interventions: Other: placebo comparator
- multiple dose 10 mg (Active Comparator): three consecutive daily intravenous injections of 10 mg DC-TAB
  Interventions: Biological: recombinant human alpha B-crystallin
- multiple dose 25 mg (Active Comparator): three consecutive daily intravenous injections of 25 mg DC-TAB
  Interventions: Biological: recombinant human alpha B-crystallin
- multiple dose 37.5 mg (Active Comparator): three consecutive daily intravenous injections of 37.5 mg DC-TAB
  Interventions: Biological: recombinant human alpha B-crystallin
- multiple dose placebo (Placebo Comparator): three consecutive daily intravenous injections of placebo
  Interventions: Other: placebo comparator

INTERVENTIONS:
Biological: recombinant human alpha B-crystallin — intravenous injection
  Other Names: HspB5; CRYAB; DC-TAB
  Arms: multiple dose 10 mg; multiple dose 25 mg; multiple dose 37.5 mg; single dose 12.5 mg; single dose 25 mg; single dose 37.5 mg; single dose 4 mg
Other: placebo comparator — intravenous injection
  Other Names: phosphate-buffered saline
  Arms: multiple dose placebo; single dose placebo

SUMMARY:
The purpose of this study is to determine safety and appropriate dose of DC-TAB for selective immune tolerance induction in humans.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, placebo-controlled, dose-escalation study of DC-TAB in healthy human volunteers. DC-TAB is a solution of the small heat-shock protein alpha B-crystallin for intravenous injection, designed to induce selective immunological tolerance as a treatment for multiple sclerosis. In this first-in-man study, DC-TAB is administered to healthy subjects in varying doses and for a varying number of times, after which safety and tolerability is evaluated, as well as the impact of the treatment on antigen-specific responses by peripheral blood T cells and serum antibodies. Blood samples are additionally collected to measure serum concentrations of DC-TAB, and to determine the rate of clearance from the circulation. The study is double blind and placebo-controlled to strengthen the significance especially of immunological evaluations.

The study consists of two parts. In Part 1, subjects receive a single dose of DC-TAB or placebo whereas in Part 2, (different) subjects receive DC-TAB or placebo on 3 consecutive days. In Part 1, four groups of subjects (n=10) are studied in a single dose, dose-escalation design. Each group of subjects are randomized to receive either DC-TAB (n=8) or placebo (n=2) once. In Part 2, three groups of subjects (n=12) are studied in a multiple dose, dose-escalation design. Each group of subjects are randomized to receive either DC-TAB (n=9) or placebo (n=3) once daily on 3 consecutive days. The next higher dose group in each part of the study only starts once safety data up to 4 days for Part 1, up to 8 days for Part 2 of the previous dose group have been reviewed and have raised no safety concerns. Part 2 is started once all safety data of Part 1 have been reviewed. Immunological effects of the treatments are evaluated over a period of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Signed the written informed consent form before first screening procedure
* Age ≥ 18 years and ≤ 55 years
* In general good health in the opinion of the investigator
* BMI between 20.0 and 28.0 kg/m2
* Use of adequate and stable contraception for 3 months prior to study initiation, during the course of the study and 30 days thereafter. Sexually active males must use a condom. Sexually active females must use double-barrier contraception or hormonal contraceptive (oral, transdermal, vaginal ring, implants), or must have undergone clinically documented total hysterectomy and/or oophorectomy, surgical sterilization or be postmenopausal defined by amenorrhea for at least 12 months and confirmed with a FSH higher than 40 IU/mL.
* If subjects claim abstinence as their method of contraception, they must be willing to agree to use condoms if they become sexually active from 14 days prior to the first dose of the study drug through 90 days beyond the conclusion of the study.

Exclusion Criteria:

* Pregnant women, women planning to become pregnant and breastfeeding women
* Subjects with a history of MS in first grade family members
* A history of or currently active clinically significant cardiac (including clinically significant ECG abnormalities in the opinion of the PI), pulmonary, gastrointestinal, hepatic, renal, pancreatic, or neurological disease
* ALT, AST and/or gamma-GT above 3 times the upper limit of normal
* Serum creatinine above 1.5 times the upper limit of normal
* Amylase above 1.5 times the upper limit of normal
* Hemoglobin < 7.0 mmol/L for females and < 8 mmol/L for males; leucocytes > 20*109/L or < 3.5*109/L; platelets < 125*109/L
* SBP > 160 mmHg and/or DBP > 100 mmHg
* Known or suspected hypersensitivity to any component of DC-TAB
* Known or suspected impairment of the immune system
* Acute respiratory or other active infections or illnesses
* Fever (oral temperature > 38.0 °C on day 1)
* Blood donation or significant blood loss within 90 days of first study medication dosing.
* Plasma donation within 7 days of first study medication dosing
* Recipients of blood or blood products in the last 6 months
* Participation in another clinical study within 90 days of the start of this trial or planning participation in another clinical trial during this study or in the 4 weeks after last visit
* Taking immunosuppressive agents, corticosteroids, anti-allergic, anti-coagulation or anti-platelet medication
* History of drug addiction (positive drug screen) or excessive use of alcohol (weekly intake more than 28 units of alcohol), or psychological or other emotional problems that are likely to invalidate informed consent, or limit the ability of the subject to comply with the protocol requirements
* Positive HIV1, or HIV2 serology
* Positive results from the hepatitis serology which indicates acute or chronic hepatitis B or hepatitis C
* Positive alcohol breath test
* Vaccination with any vaccine within 4 weeks prior to dosing of the study medication
* Any physical condition that would, in the opinion of the investigator, place the subject at an unacceptable health risk or risk of injury or render the subject unable to meet the requirements of the protocol
* History of serious adverse reactions or hypersensitivity to any medicinal product
* Smoking > 5 cigarettes/day or unable to refrain from smoking while confined to the CPU
* Use of prescription, over-the-counter (OTC), herbal supplements (excluding hormonal contraceptives, one-a-day vitamins, acetaminophen) within 14 days prior to the first dose of study drug).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events) | 28 days
  Frequency of

SECONDARY OUTCOMES:
Antigen-specific T-cell response | 28 days
  Strength of antigen-specific T-cell responses
Pharmacokinetics (serum levels of DC-TAB) | 24 h
  Serum levels of DC-TAB
Local tolerability (Injection site abnormalities) | 28 days
  Injection site abnormalities
Antibody responses | 28 days
  Serum levels of anti-DC-TAB antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Floris Höppener, PhD, MD, Principal Investigator — Syneos Health
Locations (1):
- Kendle International, Utrecht, Netherlands

REFERENCES:
- [Derived] van Noort JM, Bsibsi M, Nacken PJ, Verbeek R, Venneker EH. Therapeutic Intervention in Multiple Sclerosis with Alpha B-Crystallin: A Randomized Controlled Phase IIa Trial. PLoS One. 2015 Nov 23;10(11):e0143366. doi: 10.1371/journal.pone.0143366. eCollection 2015. PMID 26599332